CLINICAL TRIAL: NCT00135577
Title: A Double-Blind, Placebo-Controlled, Multicenter Phase IIb Extension Study to Evaluate the Safety and Efficacy of Multiple Alvimopan Dosage Regimens for the Treatment of Opioid-Induced Bowel Dysfunction in Cancer Pain Subjects
Brief Title: Study 767905/008 Extension Study: Alvimopan for Treatment of Opioid-Induced Bowel Dysfunction in Cancer Pain Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABD101684
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2009-09

CONDITIONS: Cancer; Bowel Dysfunction
Keywords: opioids; constipation; opioid-induced bowel dysfunction
MeSH Terms: conditions — Neoplasms; Intestinal Diseases; Constipation; Opioid-Induced Constipation | interventions — alvimopan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Alvimopan 0.5 mg Twice Daily (BID) (Experimental): 0.5 milligrams (mg) of alvimopan was administered orally once in the morning and once in the evening.
  Interventions: Drug: alvimopan
- Alvimopan 1 mg Once Daily (QD) (Experimental): Participants who did not have an interruption in blinded investigational product between the original study and the extension study received Alvimopan 1 mg in the morning and received placebo in the evening.
  Participants who had an interruption in blinded investigational product between studies received 0.5 mg of alvimopan in the morning and placebo in the evening for 3 days, then 1 mg of alvimopan in the morning and placebo in the evening for the remaining 3 weeks.
  Interventions: Drug: alvimopan; Drug: placebo
- Alvimopan 1 mg Twice Daily (BID) (Experimental): Participants who did not have an interruption in blinded investigational product between the original study and the extension study received Alvimopan 1 mg once in the morning and once in the evening.
  Participants who had an interruption in blinded investigational product between studies received 0.5 mg of alvimopan once in the morning and once in the evening for 3 days, then 1 mg of alvimopan once in the morning and once in the evening.
  Interventions: Drug: alvimopan
- Placebo (Placebo Comparator): Placebo was administered orally once in the morning and once in evening.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: alvimopan
  Arms: Alvimopan 0.5 mg Twice Daily (BID); Alvimopan 1 mg Once Daily (QD); Alvimopan 1 mg Twice Daily (BID)
Drug: placebo
  Arms: Alvimopan 1 mg Once Daily (QD); Placebo

SUMMARY:
Study SB-767905/008 was a multicenter study to evaluate the effectiveness and safety of multiple dosage regimens of an investigational drug for the treatment of constipation due to prescription pain medication in participants with cancer pain.

Study ABD101684 will serve as an extension to Study SB-767905/008 and offer continued access to blinded investigational product to participants who have completed the original study. The purpose of Study ABD101684 is to evaluate the safety and efficacy of alvimopan compared to placebo in subjects who completed Study SB-767905/008 and elected to participate in this extension study.

ELIGIBILITY:
Inclusion Criteria:

* Completed GSK sponsored alvimopan (opioid-induced bowel dysfunction) OBD study for subjects with cancer-related pain, e.g. SB-767905/008.
* Taking full agonist opioid therapy for cancer related pain.
* Met entry criteria of OBD in original study and per investigator continues to require therapy for management of OBD.
* Capable of completing paper questionnaires at the study visits.

Exclusion Criteria:

* Unable to eat or drink.
* Taking opioids for management of drug addiction.
* Unable to use only rescue laxatives provided.
* Inappropriately managed severe constipation that puts subject at risk of complications.
* Has gastrointestinal (GI) or pelvic disorder known to affect bowel transit.
* Concomitant medication(s), medical condition, or clinically significant laboratory abnormality that could jeopardize subject and also contraindicate study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2004-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Incidence of reported adverse events, including serious adverse events

SECONDARY OUTCOMES:
Incidence of treatment-limiting toxicities, changes in pain intensity, patient satisfaction, health outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (39):
- United States (14):
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, La Verne, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Des Moines, Iowa
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Hendersonville, North Carolina
  - GSK Investigational Site, Tacoma, Washington
- Canada (7):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, Bonaventure, Quebec
  - GSK Investigational Site, Chandler, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- GSK Investigational Site, Helsinki, Finland
- France (4):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Vandœuvre-lès-Nancy
  - GSK Investigational Site, Villejuif
- GSK Investigational Site, Kwun Tong, Hong Kong
- GSK Investigational Site, Wellington, New Zealand
- GSK Investigational Site, Lahore, Pakistan
- GSK Investigational Site, Lima, Lima Province, Peru
- Poland (5):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Otwock
  - GSK Investigational Site, Poznan
- GSK Investigational Site, Lisbon, Portugal
- GSK Investigational Site, Moscow, Russia
- GSK Investigational Site, Alcorcón, Spain
- GSK Investigational Site, Nottingham, United Kingdom